CLINICAL TRIAL: NCT06292377
Title: Better Understanding of Fatigue After STroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of Neurology Department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BRUFAST
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Electrocardiography; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients (Experimental): Patients, hospitalized at the Stroke Unit of CHU Brugmann and UZ Brussel, after the clinical diagnosis of a first-ever ischemic stroke.
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Transthoracic echography (TTE); Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: ECG — An electrocardiogram (ECG) is a simple, non-invasive test that records the electrical activity of the heart.
Diagnostic Test: Transthoracic echography (TTE) — A transthoracic echocardiogram (TTE) is a test that uses ultrasound (sound waves) to create images of the heart.
Diagnostic Test: Blood sampling — Blood sampling will include: complete blood count, serum creatinine and electrolytes, liver enzymes, fast lipid profile, glucose, HbA1C, thyroid-stimulating hormone (TSH), CRP, iron status, cardiac troponin (cTnT), N-terminal pro-brain natriuretic peptide (NT-proBNP).

SUMMARY:
Stroke is worldwide the second most common cause of death following heart attack and the leading cause of disability. Post-stroke fatigue (PSF) is a common complication after stroke and can be defined as 'an overwhelming exhaustion or tiredness, not related to exertion, which does not typically improve with rest'. Fatigue following stroke can be divided into early (< 3 months) and late (> 3 months) fatigue. PSF can have a considerable impact on a person's everyday activities and quality of life, participation in the rehabilitation process and levels of caregiver burden. Yet no efficient treatment exists to prevent or cure PSF because the pathophysiology remains unclear and seems to be multifaceted.

Autonomic dysfunction is a common complication after stroke, associated with higher morbidity and mortality. An easy tool to measure the function of the autonomic nervous system (ANS) is heart rate variability (HRV), which is defined as the beat-to-beat variation of the heart rate (= interbeat interval (IBI)). It is the result of alterations in the sympathetic and parasympathetic nervous system. In recent systematic reviews, authors stipulate that HRV can be regarded as a prognostic factor for short- and long-term stroke outcomes. HRV can be derived from 24 hours, 5 minutes (short-term) and < 5 minutes (ultra-short-term) measurements by applying time-domain and frequency-domain indices.

Autonomic dysfunction has been related to chronic fatigue syndrome, in addition to fatigue in multiple sclerosis, Parkinson's disease and myasthenia gravis. However, to the best of our knowledge, the relationship between autonomic dysfunction and PSF has not yet been fully investigated.

Fatigue is also common in cardiovascular diseases, especially in patients with heart failure (HF). HF can contribute to fatigue after stroke, independently of stroke.

Cardiac complications after acute ischemic stroke (AIS), such as arrhythmias, cardiac dysfunction and myocardial injury, are frequent. The so-called 'stroke-heart syndrome', a concept introduced in 2018, describes a broad spectrum of cardiac changes observed in 10-20% of patients with AIS within the first month after stroke onset, with a peak in the first 72 hours. A dysregulation in the neural-cardiac control after stroke is suspected to be the cause of the cascade leading to cardiac complications, in which autonomic dysfunction and inflammation seem to be part of the underlying mechanism.

Based on previous studies and by analogy with other neurological diseases, the investigators hypothesize that autonomic dysfunction following AIS contributes to PSF and that patients presenting heart failure as a complication following AIS have an increased risk of PSF.

To confirm this hypothesis, the investigators will conduct a prospective, interventional study where patients who are hospitalized at the Stroke Unit, within 72 hours after stroke symptom onset, will be included. Evaluation will take place of (a) the relationship between autonomic dysfunction (HRV) and early and late PSF, and of (b) the relationship between cardiac dysfunction and early PSF and late PSF.

There will also be an investigation into following elements:

* the association between early and late PSF and (a) certain inflammatory markers at admission (CRP, NLR), (b) stroke localization and (c) baseline imaging markers of brain frailty.
* the role of pre-existing fatigue + pre-existing or post-stroke newly diagnosed cognitive impairment, depression and sleep disturbances on the course of PSF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* First-ever (suspicion of) ischemic stroke based on clinical examination and/or brain imaging
* Onset < 72h at time of inclusion
* Admitted at the stroke unit of CHU Brugmann and UZ Brussel
* Ability to participate in assessment of fatigue, cognitive, mood and sleep disturbances
* Ability to undergo MRI of the brain

Exclusion Criteria:

* Unable to speak French, Dutch or English
* Pre-existing stroke or other structural brain lesion
* Life expectancy < 1 year
* Severe language impairment or dementia impeding assessment of fatigue, cognitive, mood and sleep disturbances
* Pregnancy or wish to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | Baseline (hospital admission)
  Heart rate variability is assessed by ECG monitoring and analyzed by means of Kubios software.
Heart rate variability (HRV) | 3 months after baseline
  Heart rate variability is assessed by ECG monitoring and analyzed by means of Kubios software.
Heart rate variability (HRV) | 12 months after baseline
  Heart rate variability is assessed by ECG monitoring and analyzed by means of Kubios software.
Transthoracic echography (TTE) | Baseline (hospital admission)
  Cardiac function will be evaluated by a cardiologist with transthoracic echography (TTE).
Transthoracic echography (TTE) | 3 months after baseline
  Cardiac function will be evaluated by a cardiologist with transthoracic echography (TTE).
Transthoracic echography (TTE) | 12 months after baseline
  Cardiac function will be evaluated by a cardiologist with transthoracic echography (TTE).
Fatigue Severity Scale | Baseline (hospital admission)
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a questionnaire with 9 statements rated from 1 (disagree) to 7 (agree). A total score of less than 36 suggests that the patient may not be suffering from fatigue. A total score of 36 or more suggests that the patient may need further evaluation by a physician.
Fatigue Severity Scale | 3 months after baseline
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a questionnaire with 9 statements rated from 1 (disagree) to 7 (agree). A total score of less than 36 suggests that the patient may not be suffering from fatigue. A total score of 36 or more suggests that the patient may need further evaluation by a physician.
Fatigue Severity Scale | 12 months after baseline
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a questionnaire with 9 statements rated from 1 (disagree) to 7 (agree). A total score of less than 36 suggests that the patient may not be suffering from fatigue. A total score of 36 or more suggests that the patient may need further evaluation by a physician.
N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline (hospital admission)
  NT-proBNP blood levels
N-terminal pro-brain natriuretic peptide (NT-proBNP) | 3 months after baseline
  NT-proBNP blood levels
N-terminal pro-brain natriuretic peptide (NT-proBNP) | 12 months after baseline
  NT-proBNP blood levels
cardiac troponin (cTnT) | Baseline (hospital admission)
  cardiac troponin blood levels

SECONDARY OUTCOMES:
Blood CRP level | Baseline (hospital admission)
  C-reactive protein (CRP) level in the blood (inflammatory marker)
Blood neutrophil-to-lymphocyte ratio (NLR) | Baseline (hospital admission)
  The neutrophil-to-lymphocyte ratio (NLR), calculated by dividing the neutrophil count by the lymphocyte count, is an inflammatory marker.
Stroke localization in the brain | Baseline (hospital admission)
  Manual segmentation of the acute ischemic lesion will be performed on the MRI of the brain
Fazekas scale | Baseline (hospital admission)
  The Fazekas scale is a widely used method to visually rate hyperintense white matter signal abnormalities in magnetic resonance imaging (MRI) data. It ranges from 0 (no lesions) to 3.
Global cortical atrophy scale | Baseline (hospital admission)
  Visual rating of cerebral atrophy on MRI images. Ranges from 0 (no lesions) to 39.
Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | Baseline (hospital admission)
  Short questionnaire designed to assess cognitive decline and dementia in elderly people. A score of ≥3.44 on the IQCODE indicates cognitive decline.
Presence for pre-existing fatigue (yes/no) | Baseline (hospital admission)
  Questionnaire (did you experience fatigue before you had your stroke' (yes/no))
Duration of pre-existing fatigue | Baseline (hospital admission)
  Questionnaire ('how long did you experience fatigue' (< 1 week, < 3 months, 3-6 months and > 6 months)
Patient Health Questionnaire-2 (PHQ-2) | Baseline (hospital admission)
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia (score from 0 to 6)
Patient Health Questionnaire-2 (PHQ-2) | 3 months after baseline
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia (score from 0 to 6)
Patient Health Questionnaire-2 (PHQ-2) | 12 months after baseline
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia (score from 0 to 6)
Montreal Cognitive Assessment (MoCA) questionnaire | 3 months after baseline
  Questionnaire. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
Montreal Cognitive Assessment (MoCA) score | 12 months after baseline
  Questionnaire.MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
Insomnia Severity Index (ISI) | Baseline (hospital admission)
  Insomnia will be assessed by using the Insomnia Severity Index (ISI). The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 3 months after baseline
  Insomnia will be assessed by using the Insomnia Severity Index (ISI). The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 12 months after baseline
  Insomnia will be assessed by using the Insomnia Severity Index (ISI). The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Complete blood count abnormalities: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Renal insufficiency: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Electrolyte imbalance: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Abnormal liver enzymes: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Dyslipidemia: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Diabetes: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Thyroid disorder: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results
Iron deficiency: yes/no | Baseline (hospital admission)
  Clinical decision based on the analysis of the blood sample results

CONTACTS AND LOCATIONS:
Overall Officials: Anissa Ourtani, MD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - UZ Brussel, Brussels

IPD SHARING:
Plan to Share IPD: No